CLINICAL TRIAL: NCT04668976
Title: A Pilot Protocol Evaluating Safety of the Medtronic Pump and Codman Catheter for the Delivery of Hepatic Arterial Infusion (HAI) Chemotherapy in Patients With Advanced Colorectal Carcinoma or Cholangiocarcinoma
Brief Title: A Study of the Use of the Medtronic Pump and Codman Catheter to Give Chemotherapy to Patients With Colorectal Carcinoma or Cholangiocarcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Benaroya Research Institute (Other)
Collaborators: Virginia Mason Hospital/Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRP19045
Record Dates: First submitted 2020-12-06; First posted 2020-12-16 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Colorectal Cancer; Cholangiocarcinoma
Keywords: Medtronic Pump; Codman Catheter; Hepatic Arterial Infusion (HAI); Floxuridine (FUDR); Gemcitabine; Oxaliplatin; Irinotecan (CPT-11); Fluorouracil; Leucovorin Calcium (Folinic Acid); Dexamethasone
MeSH Terms: conditions — Colorectal Neoplasms; Cholangiocarcinoma | interventions — Floxuridine; Gemcitabine; Oxaliplatin; Irinotecan; Fluorouracil; Panitumumab; Cetuximab

STUDY DESIGN:
Intervention Model Description: Pilot non- randomized safety study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Pump Therapy (Experimental): All patients will undergo surgery to have the Medtronic pump and Codman catheter placed appropriately before HAI therapy can begin.
  Interventions: Device: Medtronic pump and Codman catheter; Drug: Floxuridine (FUDR); Drug: Gemcitabine; Drug: Oxaliplatin; Drug: Irinotecan (CPT-11); Drug: Fluorouracil; Drug: Anti-EGFR (Panitumumab or Cetuximab)

INTERVENTIONS:
Device: Medtronic pump and Codman catheter — All patients will undergo surgery to have the Medtronic pump and Codman catheter placed appropriately before HAI therapy can begin.
Drug: Floxuridine (FUDR) — Please see Detailed Description.
Drug: Gemcitabine — Please see Detailed Description.
Drug: Oxaliplatin — Please see Detailed Description.
Drug: Irinotecan (CPT-11) — Please see Detailed Description.
Drug: Fluorouracil — Please see Detailed Description.
Drug: Anti-EGFR (Panitumumab or Cetuximab) — Please see Detailed Description.

SUMMARY:
This study is being done to answer the following question:

Is the combination of the Medtronic pump and the Codman catheter device a safe alternative to the C3000 Codman pump for delivering chemotherapy directly into the liver of patients with metastatic colorectal cancer or cholangiocarcinoma?

DETAILED DESCRIPTION:
Group 1 unresectable liver metastases from colorectal cancer

- Patients will receive either FOLFIRI, FOLFOX, Irinotecan or Irinotecan/oxaliplatin (anti- EGFR agent may be added to any of the systemic treatments) on Days 1 and 15 of each cycle, however initiation with systemic chemotherapy will not take place until 4 weeks post-surgery for pump placement.

Group 2 resectable liver metastases from colorectal cancer - Patients will receive either FOLFIRI, FOLFOX, Irinotecan or Irinotecan/oxaliplatin on Days 1 and 15 of each cycle, however initiation with systemic chemotherapy will not take place until 4 weeks post-surgery for pump placement.

Group 3 unresectable cholangiocarcinoma

- Patients will receive Gemcitabine (800 mg/m2 IV over 30 minutes) and Oxaliplatin (85 mg/ m2 IV over 120 minutes) or Gemcitabine (1000 mg/m2 IV over 30 minutes) alone on Days 1 and 15 of each cycle, however initiation with systemic chemotherapy will not take place until 4 weeks post-surgery for pump placement.

ELIGIBILITY:
Inclusion Criteria:

1. History of histologically confirmed colorectal adenocarcinoma metastatic to the liver with no clinically or radiographically confirmed extrahepatic disease (or) Histologically confirmed cholangiocarcinoma (Clinical or radiographic evidence of metastatic disease that has been resected is allowed, provided there is no recurrence in that area prior to protocol consent)
2. Confirmation of diagnosis must be performed at VMMC
3. Participant may have completely resected hepatic metastases without current evidence of other metastatic disease
4. Lab values ≤14 days prior to registration:

   ANC ≥ 1.0(9)/L Platelet count ≥ 75 (9)/L Creatinine ≤1.8 mg/dL AST 0 to 2x reference value ALK PHOS 0 to < 1.2 x reference value Tot Bili 0 to < 1.2 x reference value
5. Prior chemotherapy is acceptable if last dose of oxaliplatin or irinotecan is given ≥3 weeks prior to planned first dosing on this protocol. 5-FU or 5-FU leucovorin may be given ≥2 weeks prior to planned first dosing on this protocol. [Note: no chemotherapy to be given after resection of liver lesions prior to treatment on this study]
6. Any investigation agent is acceptable if administered ≥3 months before planned first dose on this protocol
7. ECOG <=1
8. Participants ≥18 years of age

Exclusion Criteria:

1. Prior radiation to the liver (prior radiation therapy to the pelvis is acceptable if competed at least 4 weeks prior to the planned first dose of treatment on protocol)
2. Colorectal cancer that is BRAF mutant or defective in mismatch repair.
3. Active infection, ascites, hepatic encephalopathy
4. Female participants who are pregnant or lactating - or planning to become pregnant within 6 months after the end of the treatment (female participants of child-bearing potential must have negative pregnancy test ≤72 hours before treatment start)
5. If in the opinion of the treating investigator a participant has any serious medical problems which may preclude receiving this type of treatment
6. Participants with current evidence of hepatitis A, B, C (i.e., active hepatitis)
7. Participants with history or known presence of primary CNS tumors, seizures not well- controlled with standard medical therapy, or history of stroke will also be excluded
8. Serious or non-healing active wound, ulcer, or bone fracture
9. History of other malignancy, except:

   1. Malignancy treated with curative intent and with no known active disease present for ≥3 years prior to registration and felt to be at low risk for recurrence by the treating physician
   2. Adequately treated non-melanomatous skin cancer or lentigo malignant without evidence of disease
   3. Adequately treated cervical carcinoma in situ without evidence of disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-11-25 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients requiring stent replacements | 1 year
Percent frequency liver toxicity | 1 year
  Alkaline phosphatase percent toxicity, Serum bilirubin percent toxicity

SECONDARY OUTCOMES:
Overall survival | 1 year
  Overall survival is defined as the time from treatment initiation till the day of death or last follow-up whichever occurs first.
Progression free survival | 1 year
  Progression free survival is defined as the time from treatment initiation till the day of progression or death whichever occurs first. Patients that are alive without progression at the end of the study will be censored.

CONTACTS AND LOCATIONS:
Overall Officials: Hagen Kennecke, MD, Principal Investigator — Virginia mason medical Center
Locations (1):
- Virginia mason medical Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No